CLINICAL TRIAL: NCT02488122
Title: Effect of the High Impact Exercise on Bone Density in Prepuberal Girls in 12 Private Schools in Bogota - Colombia During 2016 - 2017. Open Label Randomized Controlled Trial
Brief Title: Effect of the High Impact Exercise on Bone Density in Prepuberal Girls
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Because the study has not yet sponsorship.
Sponsor: Fundación Santa Fe de Bogota (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Principal Investigator, ANA KARINA SARMIENTO, ORAL AND MAXILLOFACIAL SURGEON, Fundación Santa Fe de Bogota
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: FSFBK1
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Bone Loss, Age-Related,
Keywords: Bone Mineral Density; Isometric Exercise; Bone Growth
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Impact Exercise (Experimental): weight bearing exercises, jumps, plyometric exercises
  Interventions: Other: High Impact Exercise
- Low Impact Exercise (Sham Comparator): Walking, Strength training, Cycling, Yoga.
  Interventions: Other: Low Impact Exercise

INTERVENTIONS:
Other: High Impact Exercise — In these workouts, both feet leave the ground at the same time.
  Arms: High Impact Exercise
Other: Low Impact Exercise — A workout is low-impact if at least one of your feet remains in contact with the ground at all times.
  Arms: Low Impact Exercise

SUMMARY:
Osteoporosis has become a worldwide concern an a matter of public health as osteoporosis is a major contributing factor associated with insufficiency fracture of the spine, wrist and proximal femur, and as a result, can diminish quality of life as well as increase direct and indirect healthcare costs.

The pathophysiology of osteoporosis is based on two main factors; low bone mass and age associated architectural changes within the bone, high impact exercise in childhood can improve the peak bone mass and bone architecture. The evidence suggests that bone adaptation to increased load is optimal in early puberty (Tanner stages I and II) since around 30% of total body adult bone mass is accrued during this period.

However, the optimal exercise program for increasing peak bone mineral content is still unclear. Therefore, the aim of this study is to assess if 15 minutes of high-impact exercise three times per week improve areal bone mineral density assessed by DXA of pre pubertal girls after a ten-month regimen compared to low-impact exercise. This information could highly impact the development of public health policies directed to pre pubertal girls.

ELIGIBILITY:
Inclusion Criteria:

* Girls between ages 8 to 10
* Tanner I

Exclusion Criteria:

* Precocious menarche (within the selected timeframe)
* Chronic disorders or medications known to affect bone metabolism or musculoskeletal function.
* Body Mass Index 30 or higher
* Regular vigorous physical activity (training more than 8 hours per week)

Ages: 8 Years to 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 276 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-11 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
bone mineral density (BMD) are presented for the total Body total bone mineral density | 36 weeks
  whole body whole Amount of mineral matter per square centimeter of bones.

CONTACTS AND LOCATIONS:
Overall Officials: ANA KARINA SARMIENTO, DDS, Principal Investigator — FUNDACION SANTA FE DE BOGOTA

REFERENCES:
- [Background] Bass SL, Saxon L, Daly RM, Turner CH, Robling AG, Seeman E, Stuckey S. The effect of mechanical loading on the size and shape of bone in pre-, peri-, and postpubertal girls: a study in tennis players. J Bone Miner Res. 2002 Dec;17(12):2274-80. doi: 10.1359/jbmr.2002.17.12.2274. PMID 12469922
- [Background] Sayers A, Mattocks C, Deere K, Ness A, Riddoch C, Tobias JH. Habitual levels of vigorous, but not moderate or light, physical activity is positively related to cortical bone mass in adolescents. J Clin Endocrinol Metab. 2011 May;96(5):E793-802. doi: 10.1210/jc.2010-2550. Epub 2011 Feb 16. PMID 21325463
- [Background] Hernandez CJ, Beaupre GS, Carter DR. A theoretical analysis of the relative influences of peak BMD, age-related bone loss and menopause on the development of osteoporosis. Osteoporos Int. 2003 Oct;14(10):843-7. doi: 10.1007/s00198-003-1454-8. Epub 2003 Aug 7. PMID 12904837
- [Background] Fuchs RK, Bauer JJ, Snow CM. Jumping improves hip and lumbar spine bone mass in prepubescent children: a randomized controlled trial. J Bone Miner Res. 2001 Jan;16(1):148-56. doi: 10.1359/jbmr.2001.16.1.148. PMID 11149479
- [Background] Kontulainen SA, Hughes JM, Macdonald HM, Johnston JD. The biomechanical basis of bone strength development during growth. Med Sport Sci. 2007;51:13-32. doi: 10.1159/000103002. PMID 17505117
- [Background] Rauch F, Schoenau E. Changes in bone density during childhood and adolescence: an approach based on bone's biological organization. J Bone Miner Res. 2001 Apr;16(4):597-604. doi: 10.1359/jbmr.2001.16.4.597. PMID 11315987
- [Background] Grimston SK, Willows ND, Hanley DA. Mechanical loading regime and its relationship to bone mineral density in children. Med Sci Sports Exerc. 1993 Nov;25(11):1203-10. PMID 8289606
- [Background] Witzke KA, Snow CM. Effects of plyometric jump training on bone mass in adolescent girls. Med Sci Sports Exerc. 2000 Jun;32(6):1051-7. doi: 10.1097/00005768-200006000-00003. PMID 10862529
- [Background] MacKelvie KJ, McKay HA, Petit MA, Moran O, Khan KM. Bone mineral response to a 7-month randomized controlled, school-based jumping intervention in 121 prepubertal boys: associations with ethnicity and body mass index. J Bone Miner Res. 2002 May;17(5):834-44. doi: 10.1359/jbmr.2002.17.5.834. PMID 12009014